CLINICAL TRIAL: NCT04562571
Title: Impact of a Public Commitment Charter Associated With Patient Information Leaflets on Antibiotics Prescribed by General Practitioners
Brief Title: Impact of a Communication Toolkit on Antibiotic Prescribed by General Practitioners: a Randomised Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201701939
Record Dates: First submitted 2020-07-06; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2019-09

CONDITIONS: Antibiotic Prescription
Keywords: antibiotic; antibiotic stewardship

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Charter & patient information leaflets (Experimental): A public commitment charter promoting antibiotic stewardship, signed by the general practitioner (GP) and displayed in the practice waiting room; a non-prescription pad, to be distributed to patients when an antibiotic is not needed; and a patient information leaflet to be used when antibiotics were prescribed
  Interventions: Other: Charter & patient information leaflets
- Control (No Intervention): No intervention, eligible general practitioners randomised in the control group not informed of the intervention

INTERVENTIONS:
Other: Charter & patient information leaflets — Public commitment charter, non-prescription pad, information leaflet in case of antibiotic prescription
  Arms: Charter & patient information leaflets

SUMMARY:
This study is a pragmatic, randomised, controlled, before-after interventional study conducted in one region in France in primary care. The GPs in the intervention group will receive a public commitment charter, a non prescription pad and a patient information leaflet to be used when antibiotics are prescribed, while the control group will be not aware of the intervention.

DETAILED DESCRIPTION:
Antimicrobial resistance is a major public health threat and the overuse of antibiotics contributes to its development.

In France, outpatient antibiotic use remains above the European average. Ninety percent of antibiotics are prescribed to outpatients and 70% of these are prescribed by general practitioners.

ELIGIBILITY:
Inclusion Criteria:

* working in the Lorraine region in France
* prescribing more than 25 antibiotic items per 100 patients without a chronic illness, aged 16 to 65 years
* proportion of patients treated with critical antibiotics exceeding 27% (among patients treated with antibiotics)

Exclusion Criteria:

* practicing exclusively alternative medicine, such as homeopathy or acupuncture
* GPs reaching the retirement age in the two years following the beginning of the intervention or who were not working two years before
* GPs who had already displayed a commitment charter promoting antibiotic stewardship in their practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Impact of a public commitment charter associated with patient information leaflets on antibiotic's prescription | 2 years
  prescription rate by all included GPs of all systemic antibiotics (J01 code according to the Anatomical Therapeutic Chemical - ATC - 2017 classification) between the "before" (2017-2018) and "after" (2018-2019) period using an auto regressive integrated moving average (ARIMA) model

SECONDARY OUTCOMES:
Impact of the public commitment charter associated with patient information leaflets on broad-spectrum antibiotics' prescriptions | 2 years
  prescription rates by included GPs of amoxicillin-clavulanate (J01CR02), cephalosporins (J01DD) and fluoroquinolones (J01MA) for each eligible GP between the "before" and "after" period using an auto regressive integrated moving average (ARIMA) model
Impact of the intervention on the seasonal variation of both total antibiotic use and quinolones' use | 2 years
  ratio of the [number of prescriptions of all antibiotics / quinolones during the cold-weather season (January-March and October-December)] / [number of prescriptions of all antibiotics / quinolones during the hot-weather season (April-September)] - 1 x 100 Title: Broad-spectrum antibiotics' prescriptions between the "before" and "after" period using ANOVA models
Adherence of GPs regarding the intervention: display of the public commitment charter | 1 years
  checking visually, without the GP being informed, during the opening hours of the practice, that the charter is effectively displayed in the waiting room at month 12
Adherence of GPs regarding the intervention: use patient information leaflets | 1 years
  Estimating the number of patient information leaflets distributed to patients by GPs, from the number of pads ordered from the Regional Health Insurance
Acceptability of the intervention by GPs | 1 years
  semi-structured individual interviews with a randomised sample of GPs from the intervention group and focus groups or individual interviews with patients of the included GPs, in order to assess their perceptions regarding the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Céline Pulcini, Principal Investigator — CHRU Nancy
Locations (1):
- Université de Lorraine, Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Essilini A, Le Dref G, Bocquier A, Kivits J, Welter A, Pulcini C, Thilly N; AntibioCharte scientific committee. French general practitioners' and patients' acceptability of a public commitment charter and patient information leaflets targeting unnecessary antibiotic use: a qualitative study. Antimicrob Resist Infect Control. 2022 Feb 8;11(1):32. doi: 10.1186/s13756-022-01065-3. PMID 35135624